CLINICAL TRIAL: NCT04252768
Title: AIPAC-002 (Active Immunotherapy PAClitaxel-002): A Multicentre, Phase Ib Study to Test a New Schedule of Eftilagimod Alpha (a Soluble LAG-3 Protein) as Adjunctive to Weekly Paclitaxel in Hormone Receptor-positive Metastatic Breast Carcinoma Patients
Brief Title: A Study in Hormone Receptor-positive Metastatic Breast Carcinoma Patients to Test a New Schedule of Efti (IMP321, Eftilagimod Alpha) as Adjunctive to a Weekly Treatment Regimen of Paclitaxel
Acronym: AIPAC-002
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced by other study NCT05747794
Sponsor: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P018
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — soluble LAG-3 protein, human; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eftilagimod alpha + Paclitaxel (Experimental): The chemo-immunotherapy phase consists of 6 cycles of 4 weeks each. During each cycle the subject will receive 80 mg/m2 paclitaxel intravenously on Day 1, 8 and 15 and 30 mg efti subcutaneously on Day 1 and 15 in a 28-day (4-week) cycle. Efti will always be given after paclitaxel. The maintenance phase comprises 6 visits with 4 weekly intervals; during each such visit 30 mg efti is given subcutaneosuly as monotherapy.
  Interventions: Drug: Eftilagimod Alpha; Drug: Paclitaxel

INTERVENTIONS:
Drug: Eftilagimod Alpha — The chemo-immunotherapy phase consists of 6 cycles of 4 weeks each. During each cycle the subject will receive 30 mg efti subcutaneously on Day 1 and 15 in a 28-day (4-week) cycle. Efti will always be given after paclitaxel. The maintenance phase comprises 6 visits with 4 weekly intervals; during each such visit 30 mg efti is given subcutaneosuly as monotherapy.
  Other Names: IMP321; efti
Drug: Paclitaxel — The chemo-immunotherapy phase consists of 6 cycles of 4 weeks each. During each cycle the subject will receive 80 mg/m2 paclitaxel intravenously on Day 1, 8 and 15.

SUMMARY:
This is a multicentre, multinational Phase Ib study in female HR+ MBC patients not receiving Her2-targeted therapy. Treatment consists of a chemo-immunotherapy phase followed by a maintenance phase. The chemo-immunotherapy phase consists of 6 cycles of 4 weeks each. During each cycle the subject will receive 80 mg/m2 paclitaxel intravenously on Day 1, 8 and 15 and 30 mg efti subcutaneously on Day 1 and 15 in a 28-day (4-week) cycle. Efti will always be given after paclitaxel. The maintenance phase comprises 6 visits with 4 weekly intervals; during each such visit 30 mg efti is given subcutaneously as monotherapy. A total of 24 subjects will be enrolled into the study. The primary goal of the study is safety and tolerability profile of efti in combination with weekly paclitaxel both given the same day in contrast to subsequent days as in the AIPAC trial.

DETAILED DESCRIPTION:
This is a multicentre, multinational Phase Ib study in female HR+ MBC patients not receiving Her2-targeted therapy. Treatment consists of a chemo-immunotherapy phase followed by a maintenance phase. The chemo-immunotherapy phase consists of 6 cycles of 4 weeks each. During each cycle the subject will receive 80 mg/m2 paclitaxel intravenously on Day 1, 8 and 15 and 30 mg efti subcutaneously on Day 1 and 15 in a 28-day (4-week) cycle. Efti will always be given after paclitaxel. The maintenance phase comprises 6 visits with 4 weekly intervals; during each such visit 30 mg efti is given subcutaneously as monotherapy. A total of 24 subjects will be enrolled into the study. The primary goal of the study is safety and tolerability profile of efti in combination with weekly paclitaxel both given the same day in contrast to subsequent days as in the AIPAC trial.

ELIGIBILITY:
Inclusion Criteria (selected ones):

* Metastatic oestrogen receptor positive and/or progesterone receptor positive breast adenocarcinoma, histologically proven by biopsy of the primary tumour and/or a metastasis
* Subjects who are indicated to receive first line chemotherapy with weekly paclitaxel
* ECOG performance status 0-1
* Expected survival longer than three months

Exclusion Criteria (selected ones):

* Prior chemotherapy for metastatic breast adenocarcinoma
* Disease-free interval of less than twelve months from the last dose of adjuvant chemotherapy
* Prior high-dose chemotherapy requiring hematopoietic stem cell rescue
* Inflammatory carcinoma at time of screening
* Candidate for treatment with trastuzumab (or other Her2/neu targeted agents) or endocrine based therapy according to the applicable treatment guidelines
* Systemic chemotherapy, radiation therapy or any other investigational agent within 4 weeks, endocrine therapy within 1 week or CDK4/6 inhibitors within 5 times half-life (acc. to SPC) prior to first dose of study treatment
* Symptomatic known cerebral and/or leptomeningeal metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study indication is female metastatic HER2- HR+ breast cancer
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability profile of efti in combination with weekly paclitaxel both given the same day | up to 12 month
  Severity, frequency and duration of adverse events

SECONDARY OUTCOMES:
AUC of efti given on the same day as paclitaxel | up to 12 month
  AUC after 1st injection of efti
Cmax of efti given on the same day as paclitaxel | up to 12 month
  Cmax after 1st injection of efti
Tmax of efti given on the same day as paclitaxel | up to 12 month
  Tmax after 1st injection of efti
Peripheral IFN-gamma concentration in the blood | up to 12 month
  Changes IFN-gamma concentration in course of treatment with efti
Peripheral IP-10 concentration in the blood | up to 12 month
  Changes IP-10 concentration in course of treatment with efti
Overall response rate of efti in combination with weekly paclitaxel both given the same day | up to 12 month
  Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
Median progression free survival of efti in combination with weekly paclitaxel both given the same day | up to 20 month
  The median progression free survival with the use of efti in combination with Paclitaxel
Median overall survival of efti in combination with weekly paclitaxel both given the same day | up to 20 month
  The median time frame with overall survival with the use of efti in combination with Paclitaxel
To characterise immunogenic properties of efti in combination with weekly paclitaxel both given the same day | up to 12 month
  Screen for possible ADA

IPD SHARING:
Plan to Share IPD: Undecided